CLINICAL TRIAL: NCT05440968
Title: Comparative Effectiveness of Point-of-care Glycosylated Hemoglobin Measurement (POC-A1c) vs the Current Standard Based on Oral Glucose Tolerance Test for Early Detection of Type 2 Diabetes Mellitus (DM2) in Colombia
Brief Title: Comparative Effectiveness of POC-A1c vs the Current Standard Based on OGTT for Early Detection DM2 in Colombia
Acronym: EDDIT-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Humberto Reynales MD MSc PhD (Network)
Responsible Party: Sponsor-Investigator, Humberto Reynales MD MSc PhD, Principal Investigator - MD MSc PhD, Centro de Atencion e Investigacion Medica
Organization: Centro de Atencion e Investigacion Medica (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CGIS-DM-001-18
Record Dates: First submitted 2022-06-25; First posted 2022-07-01 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Early diagnosis; Point of Care; FINDRISC; Screening; OGTT
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Disease | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - Intervention (Other): A - After randomization, participants will be offered information on healthy lifestyles according to their score on the FINDRISC questionnaire and subsequently a POC-A1c measurement + a confirmatory test order (Oral Glucose Tolerance Test)
  Interventions: Other: Point of Care - Glycated Hemoglobin (A1c); Other: Oral Glucose Tolerance Test
- B - Control (Other): B - After randomization, will be offered the same information on healthy lifestyles according to their FINDRISC score, and will receive an order to an Oral Glucose Tolerance Test.
  Interventions: Other: Oral Glucose Tolerance Test

INTERVENTIONS:
Other: Point of Care - Glycated Hemoglobin (A1c) — Test for diagnosis of Diabetes through a Point of care device
  Arms: A - Intervention
Other: Oral Glucose Tolerance Test — Routinary diagnosis diabetes test by venous blood sample

SUMMARY:
Evaluate the impact of conducting a screening questionnaire (FINDRISC) and the implementation of a point-of-care HBA1c test for those with identified risk to suffer Diabetes in ten years, to improve the proportion of patients attending for a confirmatory test ( oral glucose tolerance test ) and evaluate the impact of such a strategy to minimize type 2 diabetes outcomes.

DETAILED DESCRIPTION:
The physician explains the study´s consistency and obtains informed consent. If the patient accepts, the FINDRISC will be checked, the inclusion and exclusion criteria will be verified and the pertinent data from the patient's medical history will be recorded in a computer.

Subsequently, subjects will be included in the study and randomized into two groups. In group A (intervention) participants will be offered information on healthy lifestyles according to their score on the FINDRISC questionnaire and subsequently a POC-A1c measurement. Participants in group B (control) will be offered the same information on healthy lifestyles according to their FINDRISC score.

Additionally, all randomized participants will be invited to undergo an oral glucose tolerance test in the CAIMED allied laboratory or in the laboratory of their choice or through their health care provider with the necessary preparation recommendations for the performance of the test. For this purpose, they will be given an order that includes the date of the screening, a follow-up number and a window of time in which they should go (i.e., 30 days and with a second attempt - maximum window at 90 days).

After 30 days from the application of the screening from the delivery of the order for the OGTT, a call will be made to the randomized subjects to check the result of the OGTT if the test was taken and request its result in case it was taken, if the test was taken, it should refer the same to the center. Otherwise, the causes of loss to follow-up will be inquired not having previously performed the recommended OGTTand a new call will be made at 90 days. In patients who, if they attended the OGTT and obtained a presumptive result of diabetes (defined as an altered oral glucose tolerance test and/or altered POC - A1C test according to American Diabetes Association guidelines), a close call will be made 30 days after the test was performed to confirm whether they initiated control of their disease. For this, it will be indicated to them that they must attend a consultation by general medicine according to what is contemplated by their benefit plan administration entity, social security administrator, giving completion to the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult, aged greater than or equal to 18 years and less than or equal to 75 years.
* Understands, accepts and agrees to sign the informed consent form.
* FINDRISC greater than or equal to 12

Exclusion Criteria:

Previous diagnosis of type 1 or type 2 diabetes mellitus.

* Pregnancy or breastfeeding at the time of inclusion in the study (referred by the subject).
* History of cancer in the subject (must be in remission for 5 years).
* Known history of familiar hyperlipidemia.
* Chronic use of systemic corticosteroids (Defined as: a dose greater than 5 mg of oral prednisolone or its equivalent and/or consumption greater than one month of the same).
* Known history of hemophilia or other coagulation disorders.
* Known history of stage IV or V chronic kidney disease.
* Known history of HIV (on antiretroviral therapy).
* History of sickle cell disease
* Known history of glucose-6-phosphate dehydrogenase deficiency
* Known history of blood transfusion in the last 3 months
* Known history of erythropoietin therapy in the last 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 902 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
Attendance of patients with knowledge of their risk for diabetes type 2 to a confirmatory test, oral glucose tolerance test | up to 90 days
  Through follow up calls and report of oral glucose tolerance test, compare the attendance arm who had Point of care of A1C with the one who didn´t

SECONDARY OUTCOMES:
Number of days that determine the application of POC-A1c compared to the current recommendations from the American Academy of Diabetes (OGTT). | 30 to 90 days
  Through follow up calls and report of oral glucose tolerance test, compare the attendance arm who had Point of care of Hb1Ac with the one who didn´t
number of patients attending the confirmatory testing as adherence to their primary care physician's recommendations and clinical practice guidelines | 30 and 90 days
  Through follow up calls and report of oral glucose tolerance test, in a window stablished by 30 and 90 days. Compare the attendace arm who had Point of care of Hb1Ac with the one who didn´t
Describe the causes of non-performance of the confirmatory test throughout a brief questionnaire | up to 90 days
  Identification of predictors of non-performance or postponement of the diagnostic test within a maximum of 90 days from the initial recommendation.

CONTACTS AND LOCATIONS:
Overall Officials: Humberto Reynales, MD MSc PhD, Principal Investigator — Physician
Locations (1):
- Maria Granados, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No
there is no purpose to share participant data with third parties

REFERENCES:
- [Background] Khan MAB, Hashim MJ, King JK, Govender RD, Mustafa H, Al Kaabi J. Epidemiology of Type 2 Diabetes - Global Burden of Disease and Forecasted Trends. J Epidemiol Glob Health. 2020 Mar;10(1):107-111. doi: 10.2991/jegh.k.191028.001. PMID 32175717
- [Background] Khunti K, Gavin JR 3rd, Boulton AJM, Blickstead R, McGill M, Ceriello A, Raz I, Sadikot S, Wood DA, Cos X, Kalra S, Das AK, Espinosa Lopez C; Berlin Declaration Steering Group. The Berlin Declaration: A call to improve early actions related to type 2 diabetes. Why is primary care important? Prim Care Diabetes. 2018 Oct;12(5):383-392. doi: 10.1016/j.pcd.2018.04.003. Epub 2018 May 8. PMID 29752222
- [Background] American Diabetes Association. Standards of Medical Care in Diabetes-2022 Abridged for Primary Care Providers. Clin Diabetes. 2022 Jan;40(1):10-38. doi: 10.2337/cd22-as01. No abstract available. PMID 35221470
- [Background] Vandersmissen GJ, Godderis L. Evaluation of the Finnish Diabetes Risk Score (FINDRISC) for diabetes screening in occupational health care. Int J Occup Med Environ Health. 2015;28(3):587-91. doi: 10.13075/ijomeh.1896.00407. PMID 26190733
- [Background] Barry E, Roberts S, Oke J, Vijayaraghavan S, Normansell R, Greenhalgh T. Efficacy and effectiveness of screen and treat policies in prevention of type 2 diabetes: systematic review and meta-analysis of screening tests and interventions. BMJ. 2017 Jan 4;356:i6538. doi: 10.1136/bmj.i6538. PMID 28052845
- [Background] Barengo NC, Tuomilehto JO. How can we identify candidates at highest risk--to screen or not to screen? Herz. 2016 May;41(3):175-83. doi: 10.1007/s00059-016-4417-5. PMID 27052353
- [Background] Jani IV, Peter TF. How point-of-care testing could drive innovation in global health. N Engl J Med. 2013 Jun 13;368(24):2319-24. doi: 10.1056/NEJMsb1214197. No abstract available. PMID 23758238
- [Background] 8. Mariano Cantillo HJ, Ocampo DF, Cuello Santana KL. Uso del instrumento FINDRISK para identificar el riesgo de prediabetes y diabetes mellitus tipo 2. Revista Repertorio de Medicina y Cirugía. 2019 Oct 25;28(3):157-63.
- [Background] Barengo NC, Tamayo DC, Tono T, Tuomilehto J. A Colombian diabetes risk score for detecting undiagnosed diabetes and impaired glucose regulation. Prim Care Diabetes. 2017 Feb;11(1):86-93. doi: 10.1016/j.pcd.2016.09.004. Epub 2016 Oct 7. PMID 27727004

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT05440968/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT05440968/ICF_001.pdf